CLINICAL TRIAL: NCT03470922
Title: A Randomized, Double-Blind Phase 2/3 Study of Relatlimab Combined With Nivolumab Versus Nivolumab in Participants With Previously Untreated Metastatic or Unresectable Melanoma
Brief Title: A Study of Relatlimab Plus Nivolumab Versus Nivolumab Alone in Participants With Advanced Melanoma
Acronym: RELATIVITY-047
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA224-047; 2024-510913-13 (Other: EU CT Number)
Record Dates: First submitted 2018-03-14; First posted 2018-03-20 (Actual); Results first posted 2022-03-29 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Melanoma
Keywords: Cancer; Advanced Cancer
MeSH Terms: conditions — Melanoma; Neoplasms | interventions — relatlimab; Nivolumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Relatlimab + Nivolumab (Experimental): Combination
  Interventions: Biological: Relatlimab; Biological: Nivolumab
- Arm B: Nivolumab (Experimental): Monotherapy
  Interventions: Biological: Nivolumab

INTERVENTIONS:
Biological: Relatlimab — Specified dose on specified day
  Arms: Arm A: Relatlimab + Nivolumab
Biological: Nivolumab — Specified dose on specified days

SUMMARY:
The purpose of this study is to determine whether relatlimab in combination with nivolumab is more effective than nivolumab monotherapy in treating unresectable melanoma or melanoma that has spread.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Participants must have histologically confirmed Stage III (unresectable) or Stage IV melanoma, per the AJCC staging system
* Participants must not have had prior systemic anticancer therapy for unresectable or metastatic melanoma
* Tumor tissue from an unresectable or metastatic site of disease must be provided for biomarker analyses

Exclusion Criteria:

* Participants must not have active brain metastases or leptomeningeal metastases
* Participants must not have uveal melanoma
* Participants must not have an active, known, or suspected autoimmune disease

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 714 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2030-12-15 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (127):
- United States (22):
  - Local Institution - 0010, Tucson, Arizona
  - Local Institution - 0020, Los Angeles, California
  - Coastal Integrative Cancer Care, San Luis Obispo, California
  - Local Institution - 0116, Santa Barbara, California
  - Local Institution - 0012, Washington D.C., District of Columbia
  - Local Institution - 0013, Jacksonville, Florida
  - Local Institution - 0117, Orlando, Florida
  - Local Institution - 0007, Tampa, Florida
  - Local Institution - 0038, Atlanta, Georgia
  - Local Institution - 0016, Chicago, Illinois
  - Local Institution - 0114, Fort Wayne, Indiana
  - Local Institution - 0077, Baltimore, Maryland
  - Local Institution - 0120, Baltimore, Maryland
  - Local Institution - 0014, Boston, Massachusetts
  - Local Institution - 0134, Boston, Massachusetts
  - Local Institution - 0015, Ann Arbor, Michigan
  - Local Institution - 0009, Minneapolis, Minnesota
  - Local Institution - 0011, Rochester, Minnesota
  - Local Institution - 0018, Charlotte, North Carolina
  - Local Institution - 0019, Allentown, Pennsylvania
  - Local Institution - 0076, Dallas, Texas
  - Local Institution - 0008, Houston, Texas
- Argentina (5):
  - Local Institution - 0135, Buenos Aires, Distrito Federal
  - Local Institution - 0002, Capital Federal, Distrito Federal
  - Local Institution - 0004, Buenos Aires
  - Local Institution - 0003, Buenos Aires
  - Local Institution - 0005, Buenos Aires
- Australia (6):
  - Local Institution - 0042, North Sydney, New South Wales
  - Local Institution - 0043, Waratah, New South Wales
  - Local Institution - 0041, Greenslopes, Queensland
  - Local Institution - 0045, Southport, Queensland
  - Local Institution - 0133, Bedford Park, South Australia
  - Local Institution - 0044, Murdoch, Western Australia
- Austria (3):
  - Local Institution - 0036, Graz, Styria
  - Local Institution - 0037, Salzburg
  - Local Institution - 0035, Vienna
- Belgium (3):
  - Local Institution - 0047, Brussels
  - Local Institution - 0049, Brussels
  - Local Institution - 0048, Ghent
- Brazil (8):
  - Local Institution - 0058, Belo Horizonte, Minas Gerais
  - Local Institution - 0057, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0061, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0073, Santa Cruz do Sul, Rio Grande do Sul
  - Local Institution - 0063, São Paulo, São Paulo
  - Local Institution - 0059, Rio de Janiro
  - Local Institution - 0060, São Paulo
  - Local Institution - 0062, São Paulo
- Canada (5):
  - Local Institution - 0124, Halifax, Nova Scotia
  - Local Institution - 0068, Ottawa, Ontario
  - Local Institution - 0128, Toronto, Ontario
  - Local Institution - 0123, Montreal, Quebec
  - Local Institution - 0075, Montreal, Quebec
- Local Institution - 0001, Santiago, Santiago Metropolitan, Chile
- Colombia (2):
  - Local Institution - 0096, Medellín, Antioquia
  - Local Institution - 0095, Bogotá
- Denmark (3):
  - Local Institution - 0105, Aarhus N, Central Jutland
  - Local Institution - 0103, Herlev
  - Local Institution - 0104, Odense
- Finland (4):
  - Local Institution - 0100, Helsinki, Uusimaa
  - Local Institution - 0102, Oulu
  - Local Institution - 0119, Tampere
  - Local Institution - 0101, Turku
- France (8):
  - Local Institution - 0084, Rennes, Ille-et-Vilaine
  - Local Institution - 0079, Amiens, Somme
  - Local Institution - 0080, Bordeaux
  - Local Institution - 0085, Lille
  - Local Institution - 0081, Marseille
  - Local Institution - 0083, Paris
  - Local Institution - 0078, Pierre-Bénite
  - Local Institution - 0082, Poitiers
- Germany (13):
  - Local Institution - 0132, Heidelberg, Baden-Wurttemberg
  - Local Institution - 0131, Tübingen, Baden-Wurttemberg
  - Local Institution - 0071, Quedlinburg, Saxony-Anhalt
  - Local Institution - 0032, Buxtehude
  - Local Institution - 0029, Cologne
  - Local Institution - 0030, Erfurt
  - Local Institution - 0027, Essen
  - Local Institution - 0033, Hanover
  - Local Institution - 0074, Homburg / Saar
  - Local Institution - 0028, Lübeck
  - Local Institution - 0072, Mannheim
  - Local Institution - 0034, München
  - Local Institution - 0031, Würzburg
- Greece (2):
  - Local Institution - 0064, Athens
  - Local Institution - 0065, Thessaloniki
- Israel (3):
  - Local Institution - 0086, Haifa
  - Local Institution - 0088, Jerusalem
  - Local Institution - 0087, Ramat Gan
- Italy (6):
  - Local Institution - 0111, Turin, Piedmont
  - Local Institution - 0109, Bergamo
  - Local Institution - 0108, Milan
  - Local Institution - 0106, Napoli
  - Local Institution - 0110, Padua
  - Local Institution - 0107, Siena
- Mexico (5):
  - Local Institution - 0094, Zapopan, Jalisco
  - Local Institution - 0091, Monterrey, Nuevo León
  - Local Institution - 0093, Cancún, Quintana Roo
  - Local Institution - 0092, Mérida, Yucatán
  - Local Institution - 0129, Veracruz
- New Zealand (3):
  - Local Institution - 0090, Dunedin
  - Local Institution - 0125, Hamilton
  - Local Institution - 0089, Tauranga
- Local Institution - 0121, Oslo, Norway
- Poland (2):
  - Local Institution - 0040, Poznan
  - Local Institution - 0039, Warsaw
- Romania (4):
  - Local Institution - 0070, Cluj-Napoca, Cluj
  - Local Institution - 0066, Bucharest
  - Local Institution - 0067, Craiova
  - Local Institution - 0069, Iași
- Russia (3):
  - Local Institution - 0113, Krasnodar
  - Local Institution - 0127, Krasnoyarsk
  - Local Institution - 0112, Moscow
- Spain (6):
  - Local Institution - 0023, A Coruña
  - Local Institution - 0024, Barcelona
  - Local Institution - 0025, Barcelona
  - Local Institution - 0026, Madrid
  - Local Institution - 0021, San Sabastian Gipuzkoa
  - Local Institution - 0022, Seville
- Sweden (4):
  - Local Institution - 0098, Gothenburg
  - Local Institution - 0099, Lund
  - Local Institution - 0118, Solna
  - Local Institution - 0122, Uppsala
- United Kingdom (5):
  - Local Institution - 0052, Bristol, Avon
  - Local Institution - 0054, Glasgow, Dumfries & Galloway
  - Local Institution - 0056, Swansea, Glamorgan
  - Local Institution - 0051, London, Greater London
  - Local Institution - 0126, Inverness, Inverness-shire

REFERENCES:
- [Derived] Regan MM, Ascierto PA MD, Lipson EJ, Palaia J, Moshyk A, Selvan A, Lao CD, Atkins MB MD, McDermott DF, Potluri R, Ranjan S, Bilthare S, Long GV, Stephen Hodi F, Tawbi H, Schadendorf D. Analysis of treatment-free survival of patients with advanced melanoma receiving nivolumab as monotherapy or in combination with relatlimab in RELATIVITY-047. J Immunother Cancer. 2025 Sep 12;13(9):e012747. doi: 10.1136/jitc-2025-012747. PMID 40940136
- [Derived] Lipson EJ, Stephen Hodi F, Tawbi H, Schadendorf D, Ascierto PA, Matamala L, Gutierrez EC, Rutkowski P, Gogas HJ, Lao CD, Menezes JJ, Dalle S, Arance A, Gaudy-Marqueste C, Chen B, Jackson W, Mukherjee S, Dolfi S, Long GV. Nivolumab plus relatlimab in advanced melanoma: RELATIVITY-047 4-year update. Eur J Cancer. 2025 Jul 25;225:115547. doi: 10.1016/j.ejca.2025.115547. Epub 2025 Jun 3. PMID 40513285
- [Derived] Tawbi HA, Hodi FS, Lipson EJ, Schadendorf D, Ascierto PA, Matamala L, Castillo Gutierrez E, Rutkowski P, Gogas H, Lao CD, Janoski De Menezes J, Dalle S, Arance AM, Grob JJ, Ratto B, Rodriguez S, Mazzei A, Dolfi S, Long GV. Three-Year Overall Survival With Nivolumab Plus Relatlimab in Advanced Melanoma From RELATIVITY-047. J Clin Oncol. 2025 May;43(13):1546-1552. doi: 10.1200/JCO.24.01124. Epub 2024 Dec 13. PMID 39671533
- [Derived] Long GV, Stephen Hodi F, Lipson EJ, Schadendorf D, Ascierto PA, Matamala L, Salman P, Castillo Gutierrez E, Rutkowski P, Gogas HJ, Lao CD, Janoski De Menezes J, Dalle S, Arance A, Grob JJ, Keidel S, Shaikh A, Sobiesk AM, Dolfi S, Tawbi HA. Overall Survival and Response with Nivolumab and Relatlimab in Advanced Melanoma. NEJM Evid. 2023 Apr;2(4):EVIDoa2200239. doi: 10.1056/EVIDoa2200239. Epub 2023 Mar 22. PMID 38320023
- [Derived] Schadendorf D, Tawbi H, Lipson EJ, Stephen Hodi F, Rutkowski P, Gogas H, Lao CD, Grob JJ, Moshyk A, Lord-Bessen J, Hamilton M, Guo S, Shi L, Keidel S, Long GV. Health-related quality of life with nivolumab plus relatlimab versus nivolumab monotherapy in patients with previously untreated unresectable or metastatic melanoma: RELATIVITY-047 trial. Eur J Cancer. 2023 Jul;187:164-173. doi: 10.1016/j.ejca.2023.03.014. Epub 2023 Mar 22. PMID 37167764
- [Derived] Raschi E, Comito F, Massari F, Gelsomino F. Relatlimab and nivolumab in untreated advanced melanoma: insight into RELATIVITY. Immunotherapy. 2023 Feb;15(2):85-91. doi: 10.2217/imt-2022-0172. Epub 2023 Jan 11. PMID 36628573
- [Derived] Tawbi HA, Schadendorf D, Lipson EJ, Ascierto PA, Matamala L, Castillo Gutierrez E, Rutkowski P, Gogas HJ, Lao CD, De Menezes JJ, Dalle S, Arance A, Grob JJ, Srivastava S, Abaskharoun M, Hamilton M, Keidel S, Simonsen KL, Sobiesk AM, Li B, Hodi FS, Long GV; RELATIVITY-047 Investigators. Relatlimab and Nivolumab versus Nivolumab in Untreated Advanced Melanoma. N Engl J Med. 2022 Jan 6;386(1):24-34. doi: 10.1056/NEJMoa2109970. PMID 34986285
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT03470922.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 714 Participants were randomized and received study treatment
Groups:
- Arm A: Relatlimab + Nivolumab: Participants receive BMS-986213 (IV fixed-dose combination relatlimab/nivolumab at a 1:3 ratio) every 4 weeks (Q4W).
  For adults, dosing is relatlimab 160 mg/nivolumab 480 mg. Adolescents ≥ 40 kg will receive adult dosing; for adolescents < 40 kg, dosing is relatlimab 2 mg/kg/nivolumab 6 mg/kg.
- Arm B: Nivolumab: Participants receive Nivolumab IV monotherapy every 4 weeks (Q4W).
  Dosing for adults is 480 mg. Adolescents ≥ 40 kg will receive adult dosing; for adolescents < 40 kg, dosing is 6 mg/kg.
Period: Overall Study
Arm/Group | Arm A: Relatlimab + Nivolumab | Arm B: Nivolumab
Started | 355 | 359
Completed (Continuing in the study) | 237 | 227
Not Completed | 118 | 132
Not completed — Death | 107 | 118
Not completed — Lost to Follow-up | 5 | 5
Not completed — Participant Withdrew Consent | 4 | 9
Not completed — Other reasons | 1 | 0
Not completed — Not reported | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Relatlimab + Nivolumab | Arm B: Nivolumab | Total
Number analyzed (Participants) | 355 | 359 | 714
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (14.1) | 61.2 (14.0) | 61.2 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 153 | 298
  Male | 210 | 206 | 416
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 20 | 47
  Not Hispanic or Latino | 144 | 147 | 291
  Unknown or Not Reported | 184 | 192 | 376
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 5 | 5
  White | 342 | 348 | 690
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 13 | 5 | 18

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Progression Free Survival (PFS) is defined as the time between the date of randomization and the date of first documented tumor progression, assessed by a blinded independent central review (BICR) (per RECIST v1.1 criteria), or death due to any cause, whichever occurs first. Subjects who die without a reported progression will be considered to have progressed on the date of their death.
Time Frame: From randomization to date of first documented tumor progression or death (up to approximately 33 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Relatlimab + Nivolumab | Arm B: Nivolumab
Number analyzed (Participants) | 355 | 359
Months | 10.12 [6.37 to 15.74] | 4.63 [3.38 to 5.62]
Statistical Analysis 1: Comparison: Arm A: Relatlimab + Nivolumab vs Arm B: Nivolumab; Test type: Superiority; p = 0.0055, Log Rank; Log-rank test stratified by LAG-3 (≥ 1% vs < 1%), BRAF (mutation positive vs mutation wild-type), AJCC M-stage (M0/M1any[0] vs M1any[1]); Cox Proportional Hazard = 0.75, 95% CI 2-sided [0.62 to 0.92]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) is defined as the time between the date of randomization and the date of death due to any cause. For subjects that are alive, their survival time will be censored at the date of last contact ("last known alive date").
Time Frame: From randomization to the date of death (up to approximately 3 years)
Reporting Status: Not Posted, anticipated posting 2031-12

3. Secondary Outcome: Overall Response Rate (ORR)
Description: Objective response rate (ORR) is defined as the number of randomized subjects who achieve a best response of complete response (CR) or partial response (PR) based on BICR assessments (using RECIST v1.1 criteria).
Time Frame: From randomization up to approximately 3 years
Reporting Status: Not Posted, anticipated posting 2031-12

4. Other Pre Specified Outcome: The Number of Participants Experiencing Adverse Events (AEs)
Description: The number of participants experiencing adverse events (AEs).
  An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment.
Time Frame: From first dose to 30 days after last dose of study therapy (up to approximately 33 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Relatlimab + Nivolumab | Arm B: Nivolumab
Number analyzed (Participants) | 355 | 359
Participants | 345 | 339

5. Other Pre Specified Outcome: The Number of Participants Experiencing Serious Adverse Events (SAEs)
Description: The number of participants experiencing serious adverse events (SAEs).
  A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose: Results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is an important medical event.
Time Frame: From first dose to 30 days after last dose of study therapy (up to approximately 33 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Relatlimab + Nivolumab | Arm B: Nivolumab
Number analyzed (Participants) | 355 | 359
Participants | 121 | 105

6. Other Pre Specified Outcome: The Number of Participants Experiencing Adverse Events (AEs) Leading to Discontinuation
Description: The number of participants experiencing adverse events (AEs) leading to discontinuation.
  An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment.
Time Frame: From first dose to 30 days after last dose of study therapy (up to approximately 33 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Relatlimab + Nivolumab | Arm B: Nivolumab
Number analyzed (Participants) | 355 | 359
Participants | 69 | 41

7. Other Pre Specified Outcome: The Number of Participant Deaths in the Study
Description: The number of participant deaths in the study.
Time Frame: From first dose up to approximately 33 months
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Relatlimab + Nivolumab | Arm B: Nivolumab
Number analyzed (Participants) | 355 | 359
Participants | 108 | 119

8. Other Pre Specified Outcome: The Number of Participants Experiencing Laboratory Abnormalities in Specific Liver Tests
Description: The number of participants with clinical laboratory test abnormalities in specific liver tests based on US conventional units.
Time Frame: From first dose to 30 days after last dose of study therapy (up to approximately 33 months)
Population: All treated participants with at least one on-treatment measurement of the corresponding laboratory parameter
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Relatlimab + Nivolumab | Arm B: Nivolumab
Number analyzed (Participants) | 342 | 345
Participants
  ALT OR AST > 3XULN | 26 | 15
  ALT OR AST> 5XULN | 11 | 7
  ALT OR AST> 10XULN | 4 | 4
  ALT OR AST > 20XULN | 0 | 2
  TOTAL BILIRUBIN > 2XULN | 2 | 5
  ALP > 1.5xULN: number analyzed (Participants) | 339 | 345
  ALP > 1.5xULN | 34 | 30
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>1.5XULN IN 1 DAY | 2 | 2
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>1.5XULN IN 30 DAYS | 2 | 2
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>2XULN IN 1 DAY | 2 | 1
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>2XULN IN 30 DAYS | 2 | 1

9. Other Pre Specified Outcome: The Number of Participants Experiencing Laboratory Abnormalities in Specific Thyroid Tests
Description: The number of participants with clinical laboratory test abnormalities in specific thyroid tests based on US conventional units.
Time Frame: From first dose to 30 days after last dose of study therapy (up to approximately 33 months)
Population: All treated participants with at least one on-treatment measurement of the corresponding laboratory parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Relatlimab + Nivolumab | Arm B: Nivolumab
Number analyzed (Participants) | 328 | 333
Participants
  TSH > ULN | 106 | 106
  TSH > ULN WITH TSH <= ULN AT BASELINE: number analyzed (Participants) | 327 | 331
  TSH > ULN WITH TSH <= ULN AT BASELINE | 84 | 82
  TSH >ULN WITH ATLEAST ONE FT3/FT4 TEST VALUE <LLN: number analyzed (Participants) | 318 | 322
  TSH >ULN WITH ATLEAST ONE FT3/FT4 TEST VALUE <LLN | 63 | 48
  TSH >ULN WITH ALL OTHER FT3/FT4 TEST VALUES >= LLN: number analyzed (Participants) | 318 | 322
  TSH >ULN WITH ALL OTHER FT3/FT4 TEST VALUES >= LLN | 7 | 7
  TSH > ULN WITH FT3/FT4 TEST MISSING: number analyzed (Participants) | 318 | 322
  TSH > ULN WITH FT3/FT4 TEST MISSING | 8 | 9
  TSH < LLN | 89 | 84
  TSH <LLN WITH TSH >= LLN AT BASELINE: number analyzed (Participants) | 327 | 331
  TSH <LLN WITH TSH >= LLN AT BASELINE | 79 | 78
  TSH <LLN WITH ATLEAST ONE FT3/FT4 TEST VALUE > ULN: number analyzed (Participants) | 318 | 322
  TSH <LLN WITH ATLEAST ONE FT3/FT4 TEST VALUE > ULN | 51 | 40
  TSH <LLN WITH ALL OTHER FT3/FT4 TEST VALUES <= ULN: number analyzed (Participants) | 318 | 322
  TSH <LLN WITH ALL OTHER FT3/FT4 TEST VALUES <= ULN | 6 | 3
  TSH < LLN WITH FT3/FT4 TEST MISSING: number analyzed (Participants) | 318 | 322
  TSH < LLN WITH FT3/FT4 TEST MISSING | 11 | 7

ADVERSE EVENTS:
Time Frame: From first dose to up to 100 days post last dose (up to approximately 33 months)
Description: There was a participant in each arm that discontinued the study for reasons unrelated to death but whose deaths records were later discovered in a public search after discontinuation so were included in the All-cause mortality totals.
Arm/Group | Arm A: Relatlimab + Nivolumab | Arm B: Nivolumab
All-Cause Mortality (participants affected / at risk) | 108/355 | 119/359
Serious Adverse Events (participants affected / at risk) | 155/355 | 140/359
Other Adverse Events (participants affected / at risk) | 314/355 | 298/359
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Relatlimab + Nivolumab (N=355) | Arm B: Nivolumab (N=359)
Acquired haemophilia (Blood and lymphatic system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 5 | 4
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 4 | 2
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Heart valve incompetence (Cardiac disorders) | 0 | 1
Immune-mediated myocarditis (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 2
Myocarditis (Cardiac disorders) | 4 | 1
Palpitations (Cardiac disorders) | 1 | 0
Right ventricular dysfunction (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 2 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 5 | 0
Adrenocortical insufficiency acute (Endocrine disorders) | 1 | 0
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 1 | 0
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypophysitis (Endocrine disorders) | 1 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Lymphocytic hypophysitis (Endocrine disorders) | 1 | 0
Autoimmune uveitis (Eye disorders) | 0 | 1
Papilloedema (Eye disorders) | 0 | 1
Ulcerative keratitis (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 0 | 1
Vogt-Koyanagi-Harada disease (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Autoimmune colitis (Gastrointestinal disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 5 | 1
Constipation (Gastrointestinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 3
Gastric volvulus (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 2 | 1
Haemoperitoneum (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 3 | 1
Asthenia (General disorders) | 1 | 1
Chest pain (General disorders) | 0 | 1
Death (General disorders) | 3 | 1
Disease progression (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 1
General physical health deterioration (General disorders) | 2 | 6
Inflammation (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 0 | 2
Pyrexia (General disorders) | 3 | 5
Sudden death (General disorders) | 0 | 2
Vascular stent stenosis (General disorders) | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 2 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Immune-mediated cholangitis (Hepatobiliary disorders) | 1 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 | 1
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 | 0
Infusion related hypersensitivity reaction (Immune system disorders) | 0 | 1
Abscess soft tissue (Infections and infestations) | 1 | 0
Arthritis infective (Infections and infestations) | 1 | 0
Asymptomatic COVID-19 (Infections and infestations) | 0 | 1
Atypical pneumonia (Infections and infestations) | 1 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 3 | 3
COVID-19 pneumonia (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 1 | 2
Cytomegalovirus colitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 2 | 0
Encephalitis (Infections and infestations) | 2 | 1
Erysipelas (Infections and infestations) | 1 | 2
Febrile infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Infected seroma (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 2 | 1
Influenza (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 5 | 3
Postoperative wound infection (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 3 | 2
Septic shock (Infections and infestations) | 2 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 1
Suspected COVID-19 (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 6
Urosepsis (Infections and infestations) | 1 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 2
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 2
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Postoperative thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Spinal cord injury (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood creatine phosphokinase MB increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Lipase increased (Investigations) | 1 | 0
Liver function test increased (Investigations) | 1 | 0
Respiratory syncytial virus test positive (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Troponin T increased (Investigations) | 0 | 1
Troponin increased (Investigations) | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 3
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Autoimmune arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 2 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Clear cell sarcoma of soft tissue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 39 | 47
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Tumour inflammation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Basilar artery thrombosis (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dysdiadochokinesis (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Limbic encephalitis (Nervous system disorders) | 0 | 1
Optic neuritis (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Paraplegia (Nervous system disorders) | 1 | 0
Radiculopathy (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 2
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 3
Immune-mediated nephritis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 2 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Immune-mediated pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1
Lichen planus (Skin and subcutaneous tissue disorders) | 0 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Tumour excision (Surgical and medical procedures) | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0
Aortic thrombosis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Embolism (Vascular disorders) | 2 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1
Hypovolaemic shock (Vascular disorders) | 2 | 0
Iliac artery stenosis (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Relatlimab + Nivolumab (N=355) | Arm B: Nivolumab (N=359)
Anaemia (Blood and lymphatic system disorders) | 50 | 37
Hyperthyroidism (Endocrine disorders) | 23 | 28
Hypothyroidism (Endocrine disorders) | 58 | 47
Abdominal pain (Gastrointestinal disorders) | 31 | 31
Constipation (Gastrointestinal disorders) | 39 | 25
Diarrhoea (Gastrointestinal disorders) | 82 | 62
Dry mouth (Gastrointestinal disorders) | 28 | 18
Nausea (Gastrointestinal disorders) | 63 | 59
Vomiting (Gastrointestinal disorders) | 33 | 20
Asthenia (General disorders) | 48 | 33
Fatigue (General disorders) | 104 | 74
Influenza like illness (General disorders) | 19 | 14
Oedema peripheral (General disorders) | 26 | 21
Pyrexia (General disorders) | 44 | 33
Urinary tract infection (Infections and infestations) | 38 | 29
Infusion related reaction (Injury, poisoning and procedural complications) | 21 | 12
Alanine aminotransferase increased (Investigations) | 36 | 21
Aspartate aminotransferase increased (Investigations) | 35 | 17
Blood creatinine increased (Investigations) | 21 | 12
Troponin increased (Investigations) | 27 | 18
Weight decreased (Investigations) | 27 | 15
Decreased appetite (Metabolism and nutrition disorders) | 55 | 27
Hyperglycaemia (Metabolism and nutrition disorders) | 19 | 24
Arthralgia (Musculoskeletal and connective tissue disorders) | 84 | 54
Back pain (Musculoskeletal and connective tissue disorders) | 48 | 30
Myalgia (Musculoskeletal and connective tissue disorders) | 34 | 19
Pain in extremity (Musculoskeletal and connective tissue disorders) | 28 | 16
Dizziness (Nervous system disorders) | 21 | 24
Headache (Nervous system disorders) | 64 | 47
Paraesthesia (Nervous system disorders) | 18 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 50 | 38
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 33 | 22
Pruritus (Skin and subcutaneous tissue disorders) | 88 | 62
Rash (Skin and subcutaneous tissue disorders) | 62 | 49
Vitiligo (Skin and subcutaneous tissue disorders) | 39 | 37
Hypertension (Vascular disorders) | 21 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/22/NCT03470922/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/22/NCT03470922/SAP_001.pdf